CLINICAL TRIAL: NCT06159374
Title: Effects of Physical Training in Altered Environmental Conditions (in a Hypoxic Thermoclimatic Chamber) on Exercise Capacity and Selected Physiological Responses of the Human Body
Brief Title: Effects of Physical Training in Altered Environmental Conditions on Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MEIN 2021/DPI/229
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hypoxia, Altitude; Cold Exposure; Heat Exposure
Keywords: training; exercise; human performance; aerobic capacity; anaerobic capacity; maximal oxygen uptake; muscle power
MeSH Terms: conditions — Altitude Sickness; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (No Intervention): Control group
- normoxia-thermoneutral (Experimental): Training performed under normoxia (200 m above sea level) and thermoneutral conditions (21°C) and constant humidity (40%);
  Interventions: Other: exercise and environmental conditions
- hypoxia-thermoneutral (Experimental): Training performed under normobaric hypoxia (3000 m above sea level) and thermoneutral conditions (21°C) and constant humidity (40%);
  Interventions: Other: exercise and environmental conditions
- normoxia-heat (Experimental): training performed under normoxia (200 m above sea level) and high ambient temperature (31°C) and constant humidity (40%);
  Interventions: Other: exercise and environmental conditions
- hypoxia-heat (Experimental): training performed under normobaric hypoxia (3,000 m above sea level) and high ambient temperature (31°C) and constant humidity (40%);
  Interventions: Other: exercise and environmental conditions
- normoxia-cold (Experimental): Training performed in normoxia (200 m above sea level) and low ambient temperature (-11°C) and constant humidity (40%).
  Interventions: Other: exercise and environmental conditions
- hypoxia-cold (Experimental): training performed under normobaric hypoxia (3,000 m above sea level) and low ambient temperature (-11°C) and constant humidity (40%);
  Interventions: Other: exercise and environmental conditions
- hypoxia-heat-humidity (Experimental): training performed under normobaric hypoxia (3,000 m above sea level) and high ambient temperature (31°C) and high humidity (70%);
  Interventions: Other: exercise and environmental conditions

INTERVENTIONS:
Other: exercise and environmental conditions — Participants will perform interval training for 4 weeks in a variety of environmental conditions. There will be a measurement of aerobic and anaerobic capacity before and after the training. Before and after the first and last workout, blood will be drawn for biochemical analysis.
  Arms: hypoxia-cold; hypoxia-heat; hypoxia-heat-humidity; hypoxia-thermoneutral; normoxia-cold; normoxia-heat; normoxia-thermoneutral

SUMMARY:
The main objective of the study is to evaluate the physiological-biochemical effects of physical training under artificially altered climatic conditions (using a hypoxic thermoclimatic chamber) in particular to determine the effect of such training on exercise capacity and physiological response, including the effect of training in high-performance athletes. The study will evaluate the effects of physical training and the simultaneous application of hypoxia and heat/cold on aerobic and anaerobic capacity and the physiological response of the human body. The aim of the study is to find the most favourable environmental conditions for physical training in order to maximise physical performance.

ELIGIBILITY:
Inclusion Criteria:

absence of medical contraindications to high-intensity physical exertion. The medical examination is required (included an exercise ECG, blood tests to exclude anemia or low hemoglobin and iron concentration)

Exclusion Criteria:

any training (including hypoxia training or exposure) performed in the 6 months prior to the beginning of the intervention

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of aerobic capacity (endurance) | 7 days before training and 7-10 days after the training. Training will last 4 weeks.
  Measurement of maximal oxygen uptake and determination of ventilatory thresholds (ergospirometry)
Measurement of anaerobic capacity | 7 days before training and 7-10 days after the training. Training will last 4 weeks.
  Measurement of maximal anaerobic power (Wingate Anaerobic Test)
Blood analysis | Before (10 min) and after (3 min) the first and last training. The training will last 4 weeks and will consist of 12 workouts
  indicators of muscle damage, inflammatory markers (interleukins), oxidative stress, lactate concentration, tissue oxygenation, selected hormones (including erythropoietin) and enzymes, HIF (hypoxia inducible factor), selected vitamins, morphology (including reticulocytes), rheology and blood biochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Maciejczyk, Prof. dr, Study Director — Departament of Physiology and Biochemistry
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No